CLINICAL TRIAL: NCT00773786
Title: A Double-Blind, Crossover Study to Assess the Effects of Nebulized Brovana Added to Tiotropium on FEV1, Hyperinflation, and Exercise Endurance Capacity in COPD
Brief Title: Effect of Brovana and Tiotropium in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASRC956
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2013-12

CONDITIONS: COPD
Keywords: COPD; Bronchodilator; arformoterol; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arformoterol (Experimental): Arformoterol twice daily for 1 week via nebulizer
  Interventions: Drug: Arformoterol (Brovana)
- Placebo (Placebo Comparator): Placebo twice daily for 1 week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arformoterol (Brovana) — twice daily via nebulizer added to maintenance daily tiotropium
  Arms: Arformoterol
Drug: Placebo — Placebo twice daily for 1 week (added to maintenance tiotropium)
  Arms: Placebo

SUMMARY:
This will be a double-blind crossover trial in 20 patient with stable COPD. Data from this study will provide proof-of-concept information on whether the (anticipated) additional bronchodilator effect of Brovana added to tiotropium will lead to a meaningful improvement in the patient-centered outcome, exercise capacity. This study will only evaluate the effects of short-term (1-week) administration of Brovana. If results are positive, it would provide preliminary data for further, multicenter investigations.

DETAILED DESCRIPTION:
Hypotheses to be tested:

Brovana nebulized twice daily added to maintenance inhaled tiotropium therapy in stable COPD patients increases:

1. Forced expiratory volume in 1 second (FEV1) at peak dose effect (approximately 2 hours after AM dosing in the laboratory)
2. Resting and exercise hyperinflation at peak dose effect (inspiratory capacity (IC) at baseline and at iso-time during exercise testing; these measurements will be approximately 2 ¼ hours after AM dosing of tiotropium plus test drug.
3. Exercise treadmill endurance time at peak dose effect (approximately 2 ¼ hours after AM dosing in the laboratory)

Patients: Twenty patients will be studied

Location: Section of Pulmonary and Critical Care, St. Francis Hospital & Medical Center, Hartford, CT

Excluded drugs:

1. Anticholinergic bronchodilators other than once-daily (AM) tiotropium at standard dose
2. Long acting beta agonist bronchodilators
3. Short acting beta agonist bronchodilators must be withheld within six hours of laboratory testing

Allowed drugs:

1. Inhaled steroids
2. Oral steroids 10 mg/day or less, at stable dose for four weeks

Removal of patients from study:

1. Withdrawal of consent
2. Documented oxygen desaturation < 85% or clinically significant problems (such as angina, significant electrocardiogram (ECG) changes, etc) during any exercise testing
3. A significant adverse event
4. Protocol violation including lack of adherence

COPD exacerbations during study:

If the patient experiences a COPD exacerbation during the study which requires a change in medication or an addition of medication (such as oral steroids or antibiotics) the study will be held until stability is reached. At that time, the study will resume, beginning with new, 1-week treatment /testing corresponding to the study sequence when the exacerbation began. If the patient does not resume stability within four weeks or has a second exacerbation, the study will be terminated.

Study design: This will be a double-blind, crossover, single-site study in COPD patients who are in stable condition. All patients in study randomized to test drug by Visit 2 will have been on steady-state tiotropium therapy, off commercial long-acting beta-agonists (LABA), and using prn short-acting beta-agonists (SABA). Only acute (i.e., 1-week) effects of Brovana will be studied. SABA will be withheld from midnight before testing on each day.

Exercise testing and inspiratory capacity (IC) measurements Incremental and steady-state endurance testing will be performed on a treadmill in the Section of Pulmonary and Critical Care Medicine. The incremental test (Visit 1) will be performed to a symptom-limited maximum, with a goal to have the test duration over approximately 10 minutes. The protocol used for this will be from Porszasz et al using simultaneous increases in treadmill speed and incline, with settings based on estimated maximal workrate. Warm-up will be 1 mph at 1% grade. This will be followed at 30-second intervals by increases in speed and incline. Patients will have breath by breath measurements of expired air using our Sensormedics equipment, via a mouthpiece. IC measurements will also be measured at rest and at every minute into exercise.

Endurance tests (Visit 2, 4, 5) will be at 75% of the maximal rate determined from the initial test. For exercise capacity, duration in exercise time will be the primary outcome variable. IC will be measured at rest and at every minute during exercise.

An ECG will be performed before each exercise test, and continuous pulse oximetry will be monitored. A physician will be in attendance at each test.

Primary Efficacy Variables:

1. Change in FEV1 near peak effect (~ 2 hours of AM laboratory dosing of tiotropium plus test drug):

   1. The primary comparison will be Δ FEV1 (@ 2-hours after Tiotropium + Brovana minus pre-dose FEV1) versus Δ FEV1 (@2-hours after Tiotropium + Placebo minus pre-dose FEV1)
   2. The analysis will be performed using a repeated-measures design, PROC GLM Repeated, SAS:
2. Change in treadmill endurance time at ~75% of maximum (Δ endurance time) Brovana versus placebo: from baseline testing on tiotropium alone compared to testing on tiotropium + study drug.

   1. The primary comparison will be Δ endurance time (@ 2 ¼ hours after Tiotropium + Brovana compared to tiotropium alone
   2. The analysis will be performed using a repeated-measures design, PROC GLM Repeated, SAS
3. Change in static (resting), iso-time, and peak exercise IC measurements, which will be used as our estimates of hyperinflation; Brovana versus placebo: from baseline testing on tiotropium alone compared to testing on tiotropium + study drug.

   a. The primary co-comparisons will be: i. Δ IC at rest (static hyperinflation) (@ 2 ¼ hours after Tiotropium + Brovana compared to tiotropium alone ii. Δ IC at iso-time (static hyperinflation) (@ 2 ¼ hours after Tiotropium + Brovana compared to tiotropium alone. We are not sure what iso-time we will use, but if all patients go six minutes into exercise, we will use the six minute mark.

   b. The analyses will be performed using a repeated-measures design, PROC GLM Repeated, SAS

Sample Size Estimation The van Noord sited earlier powered their study assuming a ~ 140 mL standard deviation for paired differences in FEV1 (determined from earlier trials), a difference of ~ 50 mL, and a power of 0.90. They achieved a 150 mL (0.150 L) difference in FEV1. For our study, using a difference of 150 mL, a standard deviation of 140 mL, and a power of 0.80, 16 patients would be sufficient.

In a study by O'Donnell et al the combination of fluticasone 250 mcg / salmeterol 50 mcg was compared to salmeterol alone and placebo. Outcome variables included spirometry, lung volumes and exercise endurance time at 75% of maximal on a cycle ergometer. The average improvement (compared to placebo) in FEV1 at Day 1 (taken from graph) was about 200 mL with both the combination and salmeterol. The treatment-difference improvement in exercise endurance time with the combination was 131 ± 31 seconds (p. < 0.004), representing a 22% improvement. For salmeterol alone it was 49 ± 37 seconds. Our study would use a treadmill rather than a cycle ergometer; this will probably lead to more dyspnea-limitation than leg fatigue limitation. We predict the Δ FEV1 at two hours post dosing (compared to tiotropium alone) with Brovana + tiotropium in our study will ~ 150 mL - a Δ not too dissimilar to the O'Donnell study Δ. To detect a 90 second difference in endurance time (1/2 way between 131 seconds and 49 seconds), and assuming a standard deviation (SD) of 35 seconds, our study would be amply powered.

Study Sequence

Visit 1:

1. Informed consent obtained
2. Inclusion/exclusion criteria met
3. History and physical examination performed
4. Post-bronchodilator spirometry for inclusion criteria
5. Patient started on tiotropium, if necessary; tiotropium dispensed, if necessary
6. If necessary: long acting bronchodilators (LABA) discontinued, ipratropium discontinued
7. Levalbuterol MDI dispensed for prn use
8. Appointment given for Visit 1

Visit 2: 1 day (for patients already on tiotropium) to 1 week (those starting tiotropium) after Visit 1:

1. Brief history and limited physical
2. Spirometry on maintenance tiotropium, before AM dosing and after having SABA withheld for ~ 6 hours
3. Incremental treadmill endurance test
4. Patient instructed to continue taking tiotropium once daily in the morning (qAM) and levalbuterol MDI prn
5. Appointment for 2-week follow-up

Visit 3: 1 week after Visit 2, after maintenance tiotropium

1. Brief history and limited physical
2. Pre-bronchodilator spirometry (on maintenance tiotropium, levalbuterol withheld)
3. Tiotropium given (open label)
4. Spirometry 2 hours after tiotropium dosing
5. ECG 2 ¼ hour after tiotropium dosing
6. Endurance treadmill endurance test (including IC measurements) 2 ¼ hour after open-label tiotropium dosing
7. Nebulizer dispensed
8. Blinded Test drug # 1 dispensed (Brovana or placebo, 20 unit doses), instructions to take it via nebulizer bid, tiotropium continued qAM, levalbuterol MDI continued prn
9. Appointment for 1 week follow-up

Visit 4: 1 weeks after Visit 3, after test drug # 1

1. Brief history and limited physical
2. Pre-dosing spirometry (on maintenance tiotropium and Test Drug #1, levalbuterol withheld)
3. Tiotropium and Test Drug # 1 given
4. Spirometry 2 hours after above dosing
5. ECG 2 ¼ hour after above dosing
6. Endurance treadmill endurance test 2 ¼ hour after above dosing
7. Begin wash-out period: Tiotropium open-label plus prn levalbuterol continued; placebo given via nebulizer, to be taken bid (this part is single-blinded)
8. Appointment for 1 week follow-up

Visit 5: 1 week after Visit 4, after washout

1. Brief history and limited physical
2. Spirometry in AM
3. Blinded Test drug # 2 dispensed (Brovana or placebo, 20 unit doses), instructions to take it via nebulizer bid, tiotropium continued qAM, levalbuterol MDI continued prn
4. Appointment for 1 week follow-up

Visit 6: 1 week after Visit 5, after test drug # 2

1. Brief history and limited physical
2. Pre-dosing spirometry (on maintenance tiotropium and Test Drug #2, levalbuterol withheld)
3. Tiotropium and Test Drug #2 given
4. Spirometry 2 hours after above dosing
5. ECG 2 ¼ hour after above dosing
6. Endurance treadmill endurance test and IC measurements 2 ¼ hour after above dosing
7. Study terminated

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent (Approval by the St. Francis Hospital Institutional Review Board (IRB) will be required before study initiation)
2. Adults, age > 40 years
3. A clinical diagnosis of COPD, with spirometric confirmation: post-bronchodilator forced expiratory volume in 1 second / forced vital capacity (FEV1/FVC) ( < 0.70
4. Moderate, severe and very severe airflow limitation by GOLD criteria.
5. Clinically stable respiratory disease
6. The perceived ability to participate in pulmonary testing and exercise testing
7. COPD, stable state

Exclusion criteria:

1. Women of childbearing potential
2. Asthma
3. Supplemental oxygen use or anticipated oxygen desaturation < 85% at peak exercise (patients who desaturate below 85% on the incremental study will be excluded)
4. Co-morbidity that would interfere with the patient participating in the study, including the exercise testing. Examples include unstable cardiac disease, arthritis, psychological problems that would interfere with participation
5. An exacerbation requiring therapy or any change in maintenance COPD therapy within six weeks of testing
6. A history of a prolonged QT interval
7. Recent exacerbation of COPD

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard ZuWallack, MD, Principal Investigator — Saint Frnacis Hospital
Locations (1):
- St Francis Hospital and Medical center, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tiotropium + Arformoterol (Brovana), Then Tiotropium + Placebo: Participants first received Tiotropium + Brovana twice daily for 1 week via nebulizer. After a 1 week washout period, they received Tiotropium + placebo twice daily for 1 week.
- Placebo, Then Arformoterol (Brovana): Participants first received Tiotropium + Placebo twice daily for 1 week . After a 1 week washout period, they received Tiotropium + Brovana twice daily for 1 week via nebulizer.
Period: First Intervention (1 Week)
Arm/Group | Tiotropium + Arformoterol (Brovana), Then Tiotropium + Placebo | Placebo, Then Arformoterol (Brovana)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Tiotropium + Arformoterol (Brovana), Then Tiotropium + Placebo | Placebo, Then Arformoterol (Brovana)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Tiotropium + Arformoterol (Brovana), Then Tiotropium + Placebo | Placebo, Then Arformoterol (Brovana)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants randomized and received either Tiotropium + Brovana twice daily for 1 week or Tiotropium + placebo twice daily for 1 week.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 26 (6)
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: percent-predicted] | 53 (9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at 1 Week
Description: Change from baseline in Forced Expiratory Volume in 1 second (FEV1) after 1 week on Brovana or Placebo (measured 2 hours post dose). (Change = 1 week - baseline)
Time Frame: baseline and 1 week
Measure: Mean (Standard Error); unit: Liters
Groups:
- Brovana (Arformoterol): Participants who received Tiotropium + Brovana twice daily for 1 week via nebulizer
- Placebo: Participants who received Tiotropium + Placebo twice daily for 1 week.
Arm/Group | Brovana (Arformoterol) | Placebo
Number analyzed (Participants) | 20 | 20
Liters
  Trough to trough | 0.069 (0.048) | 0.010 (0.040)
  Peak to peak | 0.121 (0.037) | 0.023 (0.036)

2. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at 1 Week
Description: Change from baseline in Forced Vital Capacity (FVC) after 1 week on Brovana or Placebo. (Change = 1 week - baseline)
Time Frame: baseline and 1 week
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Brovana (Arformoterol) | Placebo
Number analyzed (Participants) | 10 | 10
Liters
  Trough to trough | 0120 (0.072) | 0.000 (0.091)
  Peak to peak | 0.080 (0.062) | -0.062 (0.064)

3. Secondary Outcome: Change From Baseline in Inspiratory Capacity at 1 Week
Description: Change from baseline in Inspiratory Capacity (IC) after 1 week on Brovana or Placebo (measured 2 hours post dose). (Change = 1 week - baseline).
Time Frame: baseline and 2 hours after dosing
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Brovana (Arformoterol) | Placebo
Number analyzed (Participants) | 20 | 20
Liters
  Trough to trough | 0.001 (0.898) | -0.019 (0.647)
  Peak to peak | 0.113 (0.063) | -0.004 (0.042)

ADVERSE EVENTS:
Time Frame: One week for each intervention
Description: Adverse event data was collection on all participants randomized into an intervention
Arm/Group | Arformoterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes